CLINICAL TRIAL: NCT02236455
Title: Effects of Complementary Therapies Delivered Via Mobile Technologies on Surgical Patients' Reports of Anxiety, Pain, and Self-Efficacy in Healing: A Pilot Randomized Controlled Trial in Iceland
Brief Title: Effects of Complementary Therapies Delivered Via Mobile Technologies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of San Francisco (Other)
Collaborators: Fulbright (Other)
Responsible Party: Principal Investigator, Margaret M. Hansen, Associate Professor, University of San Francisco
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: S5862
Record Dates: First submitted 2014-09-04; First posted 2014-09-10 (Estimated); Last update posted 2014-09-10 (Estimated); Status verified 2014-09

CONDITIONS: Acute Pain; Anxiety; Self Efficacy
Keywords: complementary medicine; state anxiety; acute pain; self-efficacy; surgery; medical music intervention; nature therapy; relaxation technique
MeSH Terms: conditions — Acute Pain; Anxiety Disorders | interventions — Imagery, Psychotherapy; Music Therapy; Relaxation Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Audio Relaxation technique (Experimental): Relaxation is a process that decreases the effects of stress on your mind and body. Relaxation techniques can help you cope with everyday stress and with stress related to various health problems, such as cancer and pain.
  Interventions: Behavioral: Audio Relaxation Technique
- Medical Music Intervention (Experimental): Music intervention is use to assist with relaxation and reduce stress levels in patients.
  Interventions: Behavioral: Medical Music Intervention
- Nature Therapy without Music (Experimental): Ecotherapy is the use of nature to reduce stress and to increase levels of well-being in patients.
  Interventions: Behavioral: Nature Therapy without Music
- Nature Therapy with Music (Experimental): Nature therapy videos were produced with and without music for surgical patients.
  Interventions: Behavioral: Nature Therapy with Music

INTERVENTIONS:
Behavioral: Audio Relaxation Technique — Audio relaxation technique created by an Icelandic Registered Nurse.
  Other Names: Guided Imagery
  Arms: Audio Relaxation technique
Behavioral: Medical Music Intervention — Audio recordings of non-lyrical relaxing music
  Other Names: Music Therapy
  Arms: Medical Music Intervention
Behavioral: Nature Therapy without Music — Nature videos of the mountains, desert, Icelandic scenery, and ocean were provided via iPads for surgical patients
  Other Names: Ecotherapy
  Arms: Nature Therapy without Music
Behavioral: Nature Therapy with Music — Nature videos of the mountains, forest, Icelandic landscape, and the ocean were provided via iPads for surgical patients
  Other Names: Ecotherapy with Music
  Arms: Nature Therapy with Music

SUMMARY:
The purpose of this study is to determine the effects of complementary therapies delivered via mobile technologies have a therapeutic effect on surgical patients' anxiety, pain, and self-efficacy in healing reports before, following, and at 10-day follow-up.

DETAILED DESCRIPTION:
Patients scheduled for same-day surgery (SDS) often experience state anxiety, which may result in increased perceptions of pain and lower self-efficacy in healing. Complementary therapies (CT), such as relaxation technique, massage, guided imagery, and acupuncture have been shown to benefit patients undergoing surgery. The aim of this study was to examine the effects of audio relaxation technique (ART), music intervention (MI), nature video application with music (NVAM), and nature video application without music (NVA) delivered via mobile technologies on patients' state anxiety, pain perception, and perceived self-efficacy in healing.

Methods A randomized controlled trial (RCT) involving 105 SDS patients, who were assigned to an ART (n = 25), MI (n = 25), NVAM (n = 15), NVA (n = 16), or a control group (n = 24) were assessed for state anxiety via the State Trait Anxiety Inventory (STAI), self-reported pain using the numeric rating scale (NRS), and self-efficacy with the general self-efficacy scale (GSE) four days prior to surgery, immediately prior and following the surgical intervention, and at day five post-operative.

ELIGIBILITY:
Inclusion Criteria:

* Age range 18-75-years
* English or Icelandic speaking
* Cognitively alert and oriented to person, place, time, and situation
* Intact visual and auditory senses

Exclusion Criteria:

* History of substance abuse
* Chronic pain lasting more than six months
* Use of narcotic medication for more than six months
* Major psychiatric disorders
* Taking prescribed medications for thought disorders
* Having ophthalmology and/or auditory surgery or impairments

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2012-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline state anxiety via the State Trait Anxiety Scale (STAI) | Ten days
  A randomized controlled trial (RCT) involving 105 SDS patients, who were assigned to an ART (n = 25), MI (n = 25), NVAM (n = 15), NVA (n = 16), or a control group (n = 24) were assessed for state anxiety via the State Trait Anxiety Inventory (STAI), self-reported pain using the numeric rating scale (NRS), and self-efficacy with the general self- efficacy scale (GSE) four days prior to surgery, immediately prior and following the surgical intervention, and at day five post-operative.

SECONDARY OUTCOMES:
Change in baseline pain level using the Numeric Rating Scale (NRS) | Ten Days
  A randomized controlled trial (RCT) involving 105 SDS patients, who were assigned to an ART (n = 25), MI (n = 25), NVAM (n = 15), NVA (n = 16), or a control group (n = 24) were assessed for state anxiety via the State Trait Anxiety Inventory (STAI), self-reported pain using the numeric rating scale (NRS), and self-efficacy with the general self- efficacy scale (GSE) four days prior to surgery, immediately prior and following the surgical intervention, and at day five post-operative.

OTHER OUTCOMES:
Change in self-efficacy in healing using the General Self-Efficacy Scale (GSE) | Ten Days
  A randomized controlled trial (RCT) involving 105 SDS patients, who were assigned to an ART (n = 25), MI (n = 25), NVAM (n = 15), NVA (n = 16), or a control group (n = 24) were assessed for state anxiety via the State Trait Anxiety Inventory (STAI), self-reported pain using the numeric rating scale (NRS), and self-efficacy with the general self- efficacy scale (GSE) four days prior to surgery, immediately prior and following the surgical intervention, and at day five post-operative.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret M Hansen, Ed.D., Principal Investigator — University of San Francisco
Locations (1):
- Landspítala, Reykjavik, Iceland

REFERENCES:
- [Result] Engwall M, Duppils GS. Music as a nursing intervention for postoperative pain: a systematic review. J Perianesth Nurs. 2009 Dec;24(6):370-83. doi: 10.1016/j.jopan.2009.10.013. PMID 19962104
- [Result] Kline GA. Does a view of nature promote relief from acute pain? J Holist Nurs. 2009 Sep;27(3):159-66. doi: 10.1177/0898010109336138. PMID 19755566
- [Result] Roykulcharoen V: The effect of a systematic relaxation technique on postoperative pain in Thailand.
- [Derived] Hansen MM. A feasibility pilot study on the use of complementary therapies delivered via mobile technologies on Icelandic surgical patients' reports of anxiety, pain, and self-efficacy in healing. BMC Complement Altern Med. 2015 Mar 28;15:92. doi: 10.1186/s12906-015-0613-8. PMID 25888344
- See also: National Center for Complementary Medicine (NIH) — http://nccam.nih.gov/